CLINICAL TRIAL: NCT05122819
Title: Evaluation of Efficacy of Intraligamentary Anesthesia by Two Different Techniques for Extraction of Mandibular Molars: A Randomized Controlled Trial
Brief Title: Evaluation of Efficacy of Intraligamentary Anesthesia for Mandibular Molar Extractions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Ayesha Basit, Associate Professor, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (21)3-4161310
Record Dates: First submitted 2021-10-14; First posted 2021-11-17 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Intraligamentary Injection by Jet Injector
  Interventions: Procedure: Mandibular Molar Extraction Under Local Anesthesia
- Group B (Experimental): Intraligamentary Injection by regular Dental Anesthesia Syringe
  Interventions: Procedure: Mandibular Molar Extraction Under Local Anesthesia
- Group C (Active Comparator): Inferior Alveolar Nerve Block
  Interventions: Procedure: Mandibular Molar Extraction Under Local Anesthesia

INTERVENTIONS:
Procedure: Mandibular Molar Extraction Under Local Anesthesia — Local Anaesthetic to be used: 2% Lidocaine in 1.8 ml cartridge (regularly used for dental anaesthesia regardless of the technique).
  Pain on injection and local anaesthesia success will be checked by using numeric pain rating scale (NPRS).

SUMMARY:
Dental extraction is the most common procedure undertaken in the department of Oral Surgery, inferior alveolar nerve block (IANB), till today, is the most commonly used local anaesthesia technique for extraction of lower posterior teeth. The anatomical complexity of this technique carries the risk of anaesthetic failures necessitating repeated needle penetrations and hence a painful experience for the patient. In addition, IANB technique, many times, becomes impossible to perform in fearful adult and paediatric patients, those with restricted mouth opening or intellectual disability. Certain coagulation defects are a contraindication to administration of IANB due to its depth of penetration into the tissues that may lead to fatal consequences in case of uncontrolled bleeding. Because of these shortcomings of IANB, there is always a need for alternative anaesthesia techniques that are less painful and carry lesser risks.

Anaesthetic injection into the Periodontal ligament space (space between tooth root surface and the bone forming the socket wall) as an alternative to IANB have been tested by many researchers with varying results. The expected advantages of this technique are reduced pain on injection, shorter duration of anaesthesia that prevents inadvertent lips and cheek biting after completion of the procedure. It is expected to be easier to perform in cases of restricted mouth opening and uncooperative patients due to any reason and carry lesser risk of bleeding within tissues.

The objective of our study is to evaluate the efficacy of Intra-ligamentary injection for posterior mandibular molar extraction as an alternative to inferior alveolar nerve block (IANB) so that it can be used in cases where IANB is either difficult to perform or not indicated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Both genders.
* Teeth selection: Mandibular first and second molars needing extraction under local anaesthesia.
* Healthy patients or those with well controlled systemic disease.
* Patients consenting to participate in the study.

Exclusion criteria:

* Patients younger than 18 years.
* Mandibular third molars, acutely inflamed or infected first and second molars.
* Pregnant patients and those with poorly controlled systemic disease.
* Mentally handicapped patients.
* Patients not consenting to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain on injection | Immediately after local anesthesia administration regardless of the technique.
  Pain on injection will be checked by using Numeric Pain Rating Scale (NPRS). NPRS is an 11 point scale in which 0: no pain, 1-3: mild pain, 4-7: moderate pain, 8-10: worst possible pain.
Local anesthesia success | 1 minute after local anesthesia administration by intraligamentary injection regardless of the syringe used. 6 minutes after administration of Inferior Alveolar Nerve Block (IANB).
  Local anesthesia success will be checked by using Numeric Pain Rating Scale (NPRS).
  NPRS is an 11 point scale in which 0: no pain, 1-3: mild pain, 4-7: moderate pain, 8-10: worst possible pain.

SECONDARY OUTCOMES:
Successful completion of Extraction | 45 minutes from the first administration of local anesthesia injection.
  Completion of extraction within 45 minutes, without changing the intervention.
  It will be measured on the following parameters:
  1. Local anesthesia success by NPRS after first administration of Intraligamentary injection (first primary outcome measure mentioned above).
  2. Local anesthesia success by NPRS after second administration of intraligamentary injection (need to repeat the same technique).
  3. Local anesthesia failure by Intraligamentary injection administered twice (as mentioned above) and need to change the technique to conventional Inferior Alveolar Nerve Block (IANB).

CONTACTS AND LOCATIONS:
Locations (1):
- Hamdard University Dental Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No